CLINICAL TRIAL: NCT03899571
Title: Duration of Prophylactic Treatment With Oseltamivir: A Randomized Clinical Trial
Brief Title: Prophylactic Treatment With Oseltamivir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, Principal Investigator, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tamiflu 2019
Record Dates: First submitted 2019-03-31; First posted 2019-04-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 days (Active Comparator): oral oseltamivir 75 mg once daily for 5 days post-exposure
  Interventions: Drug: Oseltamivir Oral Capsule for 5 days post-exposure
- 10 days (Active Comparator): oral oseltamivir 75 mg once daily for 10 days post-exposure
  Interventions: Drug: Oseltamivir Oral Capsule for 10 days post-exposure

INTERVENTIONS:
Drug: Oseltamivir Oral Capsule for 5 days post-exposure — Patients will receive oseltamivir for 5 days after last influenza exposure.
  Arms: 5 days
Drug: Oseltamivir Oral Capsule for 10 days post-exposure — Patients will receive oseltamivir for 10 days after last influenza exposure.
  Arms: 10 days

SUMMARY:
The purpose of this study is to compare the efficacy of 5-day versus 10-day oseltamivir prophylactic treatment in patients who had been exposed to influenza.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* exposure to influenza during hospitalization
* risk factors for influenza complications
* consent for participation obtained

Exclusion Criteria:

* younger than 18 years
* hematological malignancy
* hospitalized in intensive care unit
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of influenza like illness 10 days after oseltamivir prophylactic therapy | 10 days after oseltamivir prophylactic therapy
  Experiencing influenza like illness as self assessed by a patient and/or as assessed by a medical doctor while on prophylaxis with oseltamivir and during the following 10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Lepen L, Blagus R, Veluscek M, Saletinger R, Petrovec M, Bajrovic FF, Stupica D. Five-Day vs 10-Day Postexposure Chemoprophylaxis With Oseltamivir to Prevent Hospital Transmission of Influenza: A Noninferiority Randomized Open-Label Study. Open Forum Infect Dis. 2020 Jun 19;7(8):ofaa240. doi: 10.1093/ofid/ofaa240. eCollection 2020 Aug. PMID 32766383